CLINICAL TRIAL: NCT00127595
Title: A Phase II Monocentric Study of Oxaliplatin in Combination With Gemcitabine in Patients With Advanced/Metastatic Transitional Cell Carcinoma of the Urothelial Tract
Brief Title: Oxaliplatin With Gemcitabine in Patients With Carcinoma of the Urothelial Tract
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMOX
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Last update posted 2005-08-24 (Estimated); Status verified 2005-08

CONDITIONS: Carcinoma, Transitional Cell
Keywords: carcinoma of the urothelial tract
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — gemcitabine-oxaliplatin regimen

INTERVENTIONS:
Drug: gemcitabine, oxaliplatin

SUMMARY:
This is a phase II monocentric study of oxaliplatin (Ox) in combination with gemcitabine (Gem; GEMOX) in patients (pts) with advanced/metastatic transitional cell carcinoma (TCC) of the urothelial tract.

ELIGIBILITY:
Inclusion Criteria:

* Transitional cell carcinoma
* Histologically-proven
* Locally advanced unresectable or metastatic
* With at least one measurable target
* Informed consent signed

Exclusion Criteria:

* Previous chemotherapy
* Previous radiotherapy
* Performance status >=2
* Peripheral neuropathy >=1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2002-01; Study Completion 2005-04

PRIMARY OUTCOMES:
response rate (Response Evaluation Criteria in Solid Tumors [RECIST] criteria)

SECONDARY OUTCOMES:
overall survival
disease free survival
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Christine THEODORE, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France